CLINICAL TRIAL: NCT05272540
Title: Relationship Between Degree of Hydration Measured With Bioelectrical Impedance Phase Angle Analysis, Oxidative Stress and Postoperative Complications, a Prospective Study.
Brief Title: Changes in Body Water During Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Preben Kjolhede, MD, professor, Professor, University Hospital, Linkoeping
Other Study IDs: BIA
Record Dates: First submitted 2022-02-15; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Complications; Bioelectrical Impedance; Hospital Stay; Hydration
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Day case surgery: Adult patients who are operated on as outpatients in day surgery. Treatment and care follow clinical routine. Weighing on a scales measuring bioelectrical impedance data before and after the surgery is added.
- In patient surgery: Adult patients who are operated on as inpatients in hospital care. Treatment and care follow clinical routine. Weighing on a scales measuring bioelectrical impedance data before the surgery and every morning during hospital stay is added.

SUMMARY:
Fluid is added during anesthesia and surgery to maintain and balance the dynamic hemodynamics during a surgical procedure. Excess fluid after surgery is strongly correlated with morbidity and mortality. Bioelectrical impedance analysis (BIA) measures the total body water. Increased knowledge of the degree of preoperative hydration and the perioperative course can contribute to active treatment and reduced morbidity.

Women and men ≥18 years of age who are to undergo gynecological or urological operations are included in the study. The purpose is to analyze the baseline status of the degree of hydration measured as the total body water and its components, and to monitor changes in these during a postoperative course, and to look for connections between these parameters and patient characteristics, laboratory data, type of surgery, type of anesthesia, care period and onset of postoperative symptoms and complications.

DETAILED DESCRIPTION:
Background Fluid is added during anesthesia and surgery to maintain and balance the dynamic hemodynamics during a surgical procedure. The explanation for a positive fluid balance correlating with an unfavorable postoperative course is believed to be an extracellular volume expansion. Excess fluid after surgery is strongly correlated with morbidity and mortality. Increased knowledge of the degree of preoperative hydration and the perioperative course can contribute to active treatment and reduced morbidity.

Bioelectrical impedance analysis (BIA) measures the total body water expressed as a percentage of fat-free body mass. In connection with surgery and a perioperative course, there are few studies that have examined shifts in the body's fluid content with BIA.

The purpose of the study is to analyze the baseline status of the degree of hydration measured as the total body water and its components, and to monitor changes in these during a postoperative course, and to look for connections between these parameters and patient characteristics, laboratory data, type of surgery, type of anesthesia, care period and onset of postoperative symptoms and complications.

Overall hypothesis The degree of postoperative increase in the degree of hydration correlates with postoperative symptoms and complications.

Secondary hypotheses

1. The accumulated sodium supply during the day of surgery correlates with the increase in the proportion of extracellular body water postoperative day 1.
2. The development of lymphedema in patients undergoing surgery for suspected gynecological malignancy with lymph node dissection can be detected in an early postoperative course.
3. Postoperative change in the degree of hydration correlates with the onset of postoperative symptoms and/or complications.
4. Preoperatively low lean mass index increases the risk of postoperative complications through a postoperative increase in extracellular body water.
5. Patients who are readmitted for complication after surgery have a persistently increased proportion of extracellular body water.
6. In patients after day surgery in local anesthesia and sedation that are not given IV fluid, no postoperative increase in the extracellular body water is seen.
7. In hysteroscopy and transurethral cystoscopy procedures, a change in extracellular body water is seen.
8. Body mass index does not affect the precision of the measured body water composition.

Primary end-point Degree of hydration measured by bioelectrical impedance analysis

Secondary end-points

* Patients cared for as inpatient: Postoperative symptoms, duration of hospital care, postoperative complications 8 weeks after surgery. Precision of bioimpedance analysis in test-retest measurements.
* Patients operated on in day surgery: Postoperative symptoms, time to return home, complications 8 weeks after surgery. Precision of bioimpedance analysis in test-retest measurements.

Study design The study is a prospective descriptive study.

Patients Inclusion criteria

* Women and men ≥18 years of age who are to undergo gynecological or urological operations under general anesthesia, regional anesthesia, sedation or local anesthesia
* Women and men who have given informed consent to participate in the study Exclusion criteria
* Patients with pacemakers or implanted defibrillators (ICDs)
* Pregnant women with intrauterine viable pregnancy where the pregnancy should not be terminated
* Disabled patients who can not stand on the scales
* Patients with one hand or foot missing
* Patients on dialysis due to kidney failure
* Patients who are unable to understand the meaning of the study and provide informed consent

Methods All patients who undergo planned surgery at the department of gynecology and department of urology at Linköping University Hospital for an 18-month period are screened and those who meet inclusion criteria and lack exclusion criteria are asked to participate.

The degree of hydration will be measured with bioelectrical impedance analysis by weighing the patient on the Tanita MC 780 scale systematically before and after the surgery or daily during the care period. BIA data are measured in the morning with the patient fasting and after the patient has urinated.

The study is divided into 2 parts:

Sub-study 1 - patients who are operated on as outpatients in day surgery; given local anesthetics and sedation but no IV fluid.

Sub-study 2 - patients who are operated on as inpatients in hospital care; usually under general anesthesia or under regional anesthesia and routinely receive IV fluid.

Sub-study 1 Patients who are operated in day surgery Treatment and care follow clinical routine. Weighing before and after the surgery is added.

Preoperative data: Age, American Society of Anesthesiologists (ASA) class, co-morbidity, BIA data, routine blood samples.

Peroperative data: Type of surgery, operation time, anesthesia time, type of anesthesia, sedation (type/amount), peri-operative blockade, given fluid (type/volume).

Postoperative data at the hospital: Incidence of nausea and vomiting, time to go home, BIA data and lab data (oxidative stress markers before going home; see under preoperative data) and whether the patient has been admitted to the ward.

Postoperative data after discharge: Complications 8 weeks after surgery via medical record review and the Gynop register or ward nurse who calls the patient and interviews.

Sub-study 2: Patients who are operated as inpatients Treatment and care follow clinical routine. Preoperative data: Age, co-morbidity ASA class, BIA data, routine blood samples.

Clinical data: Type of surgery, operation time, anesthesia time, type of anesthesia, peroperative bleeding, urine production, given fluid (type/volume).

Postoperative data in hospital: Incidence of nausea and vomiting, BIA data, daily routine blood tests. Complications during care.

Postoperative data after discharge: Complications 8 weeks after surgery via medical examination and the Gynop register or ward nurse who calls the patient and interviews.

BIA data To validate BIA data, the first 100 patients from each sub-study and department will perform double measurements in immediate time sequence.

Lymfoedeoma Quality of Life (LYMQOL) questionnaire All participants fill in the questionnaire about "swollen legs", LYMQOL, before surgery and after 4-6 weeks and 6 months postoperatively.

Statistical considerations/power calculation No formal power calculation has been made because the study is descriptive and hypothesis-generating /exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥18 years of age who are to undergo gynecological or urological operations under general anesthesia, regional anesthesia, sedation or local anesthesia
* Women and men who have given informed consent to participate in the study

Exclusion Criteria:

* Patients with pacemakers or implanted defibrillators (ICDs)
* Pregnant women with intrauterine viable pregnancy where the pregnancy should not be terminated
* Disabled patients who can not stand on the scales
* Patients with one hand or foot missing
* Patients on dialysis due to kidney failure
* Patients who are unable to understand the meaning of the study and provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women and men ≥18 years of age who are to undergo planned gynecological or urological operations under general anesthesia, regional anesthesia, sedation or local anesthesia at the University Hospital, Linköping, Sweden.
Sampling Method: Probability Sample
Enrollment: 1696 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Perioperative change in hydration | Preoperative on day of surgery and postoperative daily during hospital stay up to 30 days after surgery
  Degree of hydration measured by bioelectrical impedance analysis

SECONDARY OUTCOMES:
Postoperative symptoms | Day of surgery until 8 week postoperatively
  Nausea, vomiting
Postoperative complications | Day of surgery until 8 week postoperatively
  According to a prespecified list of complications
Duration of hospital care | Day of surgery until 8 weeks postoperatively
  Time spent in hospital in connection with surgery either as outpatient or inpatient care
Precision of bioimpedance analysis of total body water in test-retest measurements. | Two repeated measurements preoperatively (less than 10 minutes)
  Total body water
Precision of bioimpedance analysis of intracellular water in test-retest measurements. | Two repeated measurements preoperatively (less than 10 minutes)
  Intracellular water, percent of total body water
Precision of bioimpedance analysis of extracellular water in test-retest measurements. | Two repeated measurements preoperatively (less than 10 minutes)
  Extracellular water, percent of total body water
Precision of bioimpedance analysis of phase angel in test-retest measurements. | Two repeated measurements preoperatively (less than 10 minutes)
  Phase angel, 0-90 degrees

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjölhede, Prof., Study Chair — University Hospital, Linköing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asklof M, Kjolhede P, Wodlin NB, Nilsson L. Bioelectrical impedance analysis; a new method to evaluate lymphoedema, fluid status, and tissue damage after gynaecological surgery - A systematic review. Eur J Obstet Gynecol Reprod Biol. 2018 Sep;228:111-119. doi: 10.1016/j.ejogrb.2018.06.024. Epub 2018 Jun 18. PMID 29933195